CLINICAL TRIAL: NCT07000448
Title: Effects of Personalized PEEP Titration on Postoperative Pulmonary Outcomes in Laparoscopic Hysterectomy
Brief Title: Optimal Ventilation Strategies in Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Beyhan Guner, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022-394
Record Dates: First submitted 2025-05-21; First posted 2025-06-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Recruitment Maneuver; Individualized PEEP; Total Hysterectomy; Postoperative Pulmonary Complications

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- individualized PEEP (PEEPi) (Experimental): In the patients in the PEEPᵢ group, a recruitment maneuver was performed after intubation and after the Trendelenburg position was given. The PEEP level was increased to 20 cmH₂O with 5 cmH₂O increments every five respiratory cycles, and an airway opening pressure of 40 cmH₂O was achieved. Dynamic compliance values observed on the ventilator monitor were recorded for optimal individual PEEP titration when PEEP reached 20 cmH₂O. The PEEP level was decreased by 2 cmH₂O every 3 respiratory cycles to determine the PEEP level at which the highest compliance value was achieved. 2 cmH₂O above this value was set as optimal PEEP, and this value was maintained throughout the surgery.
  Interventions: Procedure: Dynamic compliance guided individualized positive end-expiratory pressure titration strategy
- PEEP 5 (Active Comparator): Patients in the PEEP 5 group were applied a fixed 5 cmH2O PEEP, and no recruitment maneuver was performed.
  Interventions: Procedure: standardized 5 PEEP

INTERVENTIONS:
Procedure: Dynamic compliance guided individualized positive end-expiratory pressure titration strategy — For optimal individual PEEP titration, dynamic compliance values observed on the ventilator monitor were recorded when PEEP reached 20 cmH₂O.
  Arms: individualized PEEP (PEEPi)
Procedure: standardized 5 PEEP — Patients in the PEEP 5 group were applied a fixed 5 cmH2O PEEP and no recruitment maneuver was performed.
  Arms: PEEP 5

SUMMARY:
The aim of this study was to investigate whether individualized PEEP application improves respiratory function and reduces the incidence of postoperative pulmonary complications (PPCs) in patients undergoing laparoscopic total hysterectomy. Investigators hypothesized that individualized PEEP would improve pulmonary oxygenation and reduce the incidence of postoperative pulmonary complications.

DETAILED DESCRIPTION:
The study included 113 patients who met the criteria and underwent elective laparoscopic total hysterectomy.

In the patients in the PEEPᵢ group, a recruitment maneuver was performed after intubation and after the Trendelenburg position was given. During this maneuver, the ventilator was switched to pressure-controlled mode, the I:E ratio was increased to 1:1, FiO₂ was increased to 80%, and the respiratory rate was set to 15/min. The PEEP level was increased to 20 cmH₂O with 5 cmH₂O increments every 5 respiratory cycles, and an airway opening pressure of 40 cmH₂O was obtained.

For optimal individual PEEP titration, the dynamic compliance values observed on the ventilator monitor were recorded when the PEEP reached 20 cmH₂O. The PEEP level was decreased by 2 cmH₂O every 3 respiratory cycles, and the PEEP level at which the highest compliance value was obtained was determined. The value 2 cmH₂O above this value was set as optimal PEEP, and this value was maintained throughout the surgery. The recruitment maneuver was repeated at specified time points during the surgical procedure and upon disconnection of the ventilator circuit.

Data collection was performed at several time points; before induction (T1), only hemodynamic data were recorded. Before pneumoperitoneum, 5 minutes after induction (T2) with the patient in the supine position, 20 minutes after the onset of pneumoperitoneum (T3) in the Trendelenburg position, and 60 minutes after the onset of pneumoperitoneum (T4) mechanical ventilation and hemodynamic parameters were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Scheduled for elective laparoscopic total hysterectomy
* ASA physical status I-III
* BMI ≤30 kg/m²
* Anticipated surgical duration >2 hours

Exclusion Criteria:

* Pre-existing neuromuscular disorders
* NYHA class III/IV heart failure
* OSAS
* Previous lung surgery
* Severe pulmonary disease (FEV1 <50% predicted)

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 113 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Postoperative pulmonary complications (PPC) | within 7 days after surgery
  PPC included clinical conditions such as atelectasis, hypoxemia (PaO₂ < 8.0 kPa or SpO₂ < 90% on room air), pneumonia, acute respiratory distress syndrome (ARDS), pleural effusion, bronchospasm, pneumothorax, reintubation or need for non-invasive ventilation support.

SECONDARY OUTCOMES:
Intraoperative respiratory mechanics parameter | within intraoperative period
  Driving pressure
Respiratory mechanics parameter | intraoperatively
  Dynamic compliance
Mechanic ventilation parameter | during intraoperative period
  Pplatteau
Intensive care | within 7 days after surgery
  Intensive care unit (ICU) admission

CONTACTS AND LOCATIONS:
Overall Officials: Beyhan Guner, MD, Principal Investigator — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Bakirkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No